CLINICAL TRIAL: NCT04982237
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate AK104 Plus Platinum-containing Chemotherapy With or Without Bevacizumab as First-line Treatment for Persistent, Recurrent, or Metastatic Cervical Cancer
Brief Title: A Study of AK104 Plus Platinum-containing Chemotherapy±Bevacizumab as First-line Treatment for Persistent, Recurrent, or Metastatic Cervical Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK104-303
Record Dates: First submitted 2021-07-21; First posted 2021-07-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Carboplatin; Cisplatin; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104+chemotherapy± bevacizumab (Experimental): AK104 in combination with cisplatin or carboplatin and paclitaxel± bevacizumab
  Interventions: Biological: AK104; Drug: paclitaxel; Drug: carboplatin; Drug: cisplatin; Drug: bevacizumab
- Placebo+chemotherapy± bevacizumab (Placebo Comparator): Placebo in combination with cisplatin or carboplatin and paclitaxel± bevacizumab
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: cisplatin; Drug: bevacizumab; Drug: Placebo

INTERVENTIONS:
Biological: AK104 — IV infusion
  Arms: AK104+chemotherapy± bevacizumab
Drug: paclitaxel — IV infusion
Drug: carboplatin — iv infusion
Drug: cisplatin — iv infusion
Drug: bevacizumab — iv infusion
Drug: Placebo — iv infusion
  Arms: Placebo+chemotherapy± bevacizumab

SUMMARY:
This is A Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate AK104 Plus Platinum-containing Chemotherapy With or Without Bevacizumab as First-line Treatment for Persistent, Recurrent, or Metastatic Cervical Cancer

ELIGIBILITY:
Inclusion Criteria:

1. signs the written informed consent form.
2. Women aged ≥ 18 and ≤ 75 years.
3. ECOG of 0 or 1.
4. Life expectancy ≥ 3 months.
5. Histologically or cytologically confirmed cervical cancer, not amenable to curative surgery or concurrent chemoradiotherapy.

   1. The histological types include squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma;
   2. No prior systemic therapy for persistent, recurrent or metastatic ([FIGO] Stage IVB) disease.
6. At least one measurable tumor lesion per RECIST v1.1; lesions at sites previously treated with radiotherapy or other loco-regional therapy are not considered as target lesions unless the lesion has unequivocal progression or the biopsy is obtained to confirm maligancy.
7. All subjects must provide archival tumor tissue samples within 2 years prior to randomization,or fresh tumor tissue samples obtained by biopsy.
8. Subjects must have adequate organ function as assessed in the laboratory tests.
9. Female subjects of childbearing potential must have a negative serum pregnancy test prior to the first dose. If a female subject of childbearing potential must use acceptable effective methods of contraception from screening and must agree to continue these precautions until 120 days after the last dose of study drug.

Exclusion Criteria:

1. Subjects with other histopathological types of cervical cancer, such as small cell carcinoma, clear cell carcinoma, sarcoma, etc.
2. Clinically significant hydronephrosis that cannot be relieved by nephrostomy or ureteral stenting as judged by the Investigator.
3. Presence of nervous system (CNS) metastases or carcinomatous meningitis;
4. Subjects with uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
5. Patients with other active malignancies within 3 years prior to randomization.
6. Patients who have received other prior chemotherapeutic agents.
7. Any prior treatments targeting the mechanism of tumor immunity, such as anti-angiogenic therapy (e.g., bevacizumab), immune checkpoint inhibitors (e.g., anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.), or therapy against immune costimulatory factors (e.g., antibodies directed against ICOS, CD40, CD137, GITR, OX40 targets, etc).
8. Major surgical treatment, open biopsy or significant trauma within 4 weeks prior to randomization; or elective major surgical treatment required during the study.
9. Active or potentially recurrent autoimmune disease.
10. Subjects who require systemic treatment with glucocorticoid (> 10 mg/day of prednisone or equivalent glucocorticoid) or other immunosuppressive agents within 14 days prior to randomization;
11. Use of live vaccines within 4 weeks prior to randomization.
12. Known primary or secondary immunodeficiencies, including testing positive for human immunodeficiency virus (HIV) antibodies.
13. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
14. Known history of interstitial lung disease or non-infectious pneumonitis; unless induced by radiation therapies.
15. Serious infections requiring hospitalization.
16. Presence of active infection requiring systemic therapy.
17. Subjects with active hepatitis B and active viral hepatitis C.
18. Active or documented inflammatory bowel diseases, active diverticulitis.
19. Subjects with known history of severe hypersensitivity reactions to other monoclonal antibodies.
20. Known any contraindication to cisplatin/carboplatin, paclitaxel or allergy to any of their ingredients.
21. Pregnant or lactating women.
22. Any condition that, in the opinion of the Investigator, may result in a risk when receiving the study drug.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) assessed by blinded independent central review (BICR) per RECIST v1.1 | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1
overall survival (OS) | Up to approximately 2 years
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 2 years
  Proportion of subjects who have a complete or partial response relative to baseline as assessed by investigator according to RECIST 1.1 criteria
Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 2 years
  Measured from the date of partial or complete response to therapy until the cancer progresses based on RECIST v1.1 criteria.
Time to Response（TTR Per RECIST 1.1 as Assessed by BICR | Up to approximately 2 years
AE | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment
Observed concentrations of AK104 | From first dose of AK104 through 90 days after last dose of AK104
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK104 through 90 days after last dose of AK104
  The immunogenicity of AK104 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, MD, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The Second Affiliated Hospital,Anhui Medical University, Hefei
  - Fudan University Shanghai Cancer Center, Shanghai

REFERENCES:
- [Derived] Wu X, Sun Y, Yang H, Wang J, Lou H, Li D, Wang K, Zhang H, Wu T, Li Y, Wang C, Li G, Wang Y, Li D, Tang Y, Pan M, Cai H, Wang W, Yang B, Qian H, Tian Q, Yao D, Cheng Y, Wei B, Li X, Wang T, Hao M, Wang X, Wang T, Ran J, Zhu H, Zhu L, Liu X, Li Y, Chen L, Li Q, Yan X, Wang F, Cai H, Zhang Y, Liang Z, Liu F, Huang Y, Xia B, Qu P, Zhu G, Chen Y, Song K, Sun M, Chen Z, Zhou Q, Hu L, Abulizi G, Guo H, Liao S, Ye Y, Yan P, Tang Q, Sun G, Liu T, Lu D, Hu M, Wang ZM, Li B, Xia M. Cadonilimab plus platinum-based chemotherapy with or without bevacizumab as first-line treatment for persistent, recurrent, or metastatic cervical cancer (COMPASSION-16): a randomised, double-blind, placebo-controlled phase 3 trial in China. Lancet. 2024 Oct 26;404(10463):1668-1676. doi: 10.1016/S0140-6736(24)02135-4. Epub 2024 Oct 16. PMID 39426385
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39426385/